CLINICAL TRIAL: NCT04931342
Title: A Phase II, Open-Label, Multicenter, Platform Study Evaluating the Efficacy and Safety of Biomarker-Driven Therapies in Patients With Persistent or Recurrent Rare Epithelial Ovarian Tumors
Brief Title: A Study Evaluating the Efficacy and Safety of Biomarker-Driven Therapies in Patients With Persistent or Recurrent Rare Epithelial Ovarian Tumors
Acronym: BOUQUET
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: GOG Foundation (Network); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO42178; GOG-3051 (Other: GOG Foundation); ENGOT-GYN2 (Other: European Network of Gynaecological Oncological Trial Groups (ENGOT))
Record Dates: First submitted 2021-06-09; First posted 2021-06-18 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — ipatasertib; cobimetinib; Ado-Trastuzumab Emtansine; atezolizumab; Bevacizumab; Paclitaxel; giredestrant; abemaciclib; inavolisib; palbociclib; Letrozole; olaparib; Gonadotropin-Releasing Hormone; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Ipatasertib + Paclitaxel (PIK3CA/AKT1/PTEN-altered tumors) (Experimental): Participants in the Ipatasertib + Paclitaxel arm will receive treatment until unacceptable toxicity or disease progression per RECIST v1.1.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel
- Cobimetinib (BRAF/NRAS/KRAS/NF1-altered tumors) (Experimental): Participants in the Cobimetinib arm will receive treatment until unacceptable toxicity or disease progression per RECIST v1.1.
  Interventions: Drug: Cobimetinib
- Trastuzumab Emtansine (ERBB2-amplified/mutant tumors) (Experimental): Participants in the Trastuzumab Emtansine arm will receive treatment until unacceptable toxicity or disease progression per RECIST v1.1.
  Interventions: Drug: Trastuzumab Emtansine
- Atezolizumab + Bevacizumab (Non-matched) (Experimental): Participants in the Atezolizumab + Bevacizumab arm will receive treatment until unacceptable toxicity or loss of clinical benefit as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab
- Giredestrant + Abemaciclib (ER+ tumors) (Experimental): Participants in the Giredestrant + Abemaciclib arm will receive treatment until unacceptable toxicity or disease progression as determined by the investigator according to RECIST v1.1.
  Interventions: Drug: Giredestrant; Drug: Abemaciclib; Drug: Luteinizing Hormone-Releasing Hormone (LHRH) Agonists
- Inavolisib + Palbociclib (PIK3CA-altered tumors) (Experimental): Participants in the Inavolisib + Palbociclib arm will receive treatment until unacceptable toxicity or disease progression per RECIST v1.1.
  Interventions: Drug: Inavolisib; Drug: Palbociclib
- Inavolisib + Palbociclib + Letrozole (ER+ and PIK3CA-altered tumors) (Experimental): Participants in the Inavolisib + Palbociclib + Letrozole arm will receive treatment until unacceptable toxicity or disease progression per RECIST v1.1.
  Interventions: Drug: Inavolisib; Drug: Palbociclib; Drug: Letrozole; Drug: Luteinizing Hormone-Releasing Hormone (LHRH) Agonists
- Inavolisib + Olaparib (Non-matched) (Experimental): Participants in the Inavolisib + Olaparib arm will receive treatment until unacceptable toxicity or disease progression per RECIST v1.1.
  Interventions: Drug: Inavolisib; Drug: Olaparib
- Inavolisib + Giredestrant (ER+ and PIK3CA-altered tumors) (Experimental): Participants in the Inavolisib + Giredestrant arm will receive treatment until unacceptable toxicity or disease progression per RECIST v1.1.
  Interventions: Drug: Giredestrant; Drug: Inavolisib
- Inavolisib + Bevacizumab (PIK3CA-altered tumors) (Experimental): Participants in the Inavolisib + Bevacizumab arm will receive treatment until unacceptable toxicity or disease progression per RECIST v1.1.
  Interventions: Drug: Bevacizumab; Drug: Inavolisib
- Atezolizumab + Bevacizumab + Cyclophosphamide (Non-matched) (Experimental): Participants in the Atezolizumab + Bevacizumab + Cyclophosphamide arm will receive treatment until unacceptable toxicity or loss of clinical benefit as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Ipatasertib — Ipatasertib will be administered by mouth once a day on Days 1-21 of each cycle. (Cycle length = 28 days)
  Other Names: RO5532961
  Arms: Ipatasertib + Paclitaxel (PIK3CA/AKT1/PTEN-altered tumors)
Drug: Cobimetinib — Cobimetinib will be administered by mouth once a day on Days 1-21 of each cycle. (Cycle length=28 days)
  Other Names: RO5514041
  Arms: Cobimetinib (BRAF/NRAS/KRAS/NF1-altered tumors)
Drug: Trastuzumab Emtansine — Trastuzumab Emtansine will be administered intravenously on Day 1 of each cycle. (Cycle length=21 days)
  Other Names: RO5304020
  Arms: Trastuzumab Emtansine (ERBB2-amplified/mutant tumors)
Drug: Atezolizumab — Atezolizumab will be administered intravenously on Day 1 of each cycle. (Cycle length=21 days)
  Other Names: RO5541267, Tecentriq
  Arms: Atezolizumab + Bevacizumab (Non-matched); Atezolizumab + Bevacizumab + Cyclophosphamide (Non-matched)
Drug: Bevacizumab — Bevacizumab will be administered intravenously on Day 1 of each cycle. (Cycle length=21 days)
  Other Names: RO4876646, Avastin
  Arms: Atezolizumab + Bevacizumab (Non-matched); Atezolizumab + Bevacizumab + Cyclophosphamide (Non-matched); Inavolisib + Bevacizumab (PIK3CA-altered tumors)
Drug: Paclitaxel — Paclitaxel will be administered intravenously on Days 1, 8, and 15 of each cycle. (Cycle length=28 days)
  Arms: Ipatasertib + Paclitaxel (PIK3CA/AKT1/PTEN-altered tumors)
Drug: Giredestrant — Giredestrant will be administered by mouth once a day on Days 1-28 of each cycle (Cycle length=28 days)
  Arms: Giredestrant + Abemaciclib (ER+ tumors); Inavolisib + Giredestrant (ER+ and PIK3CA-altered tumors)
Drug: Abemaciclib — Abemaciclib will be administered by mouth twice a day during each 28-day cycle
  Arms: Giredestrant + Abemaciclib (ER+ tumors)
Drug: Inavolisib — Inavolisib will be administered by mouth once a day on Days 1-28 of each 28-day cycle
  Arms: Inavolisib + Giredestrant (ER+ and PIK3CA-altered tumors); Inavolisib + Olaparib (Non-matched); Inavolisib + Palbociclib (PIK3CA-altered tumors); Inavolisib + Palbociclib + Letrozole (ER+ and PIK3CA-altered tumors)
Drug: Palbociclib — Palbociclib will be administered by mouth once a day on Days 1-21 of each 28-day cycle
  Arms: Inavolisib + Palbociclib (PIK3CA-altered tumors); Inavolisib + Palbociclib + Letrozole (ER+ and PIK3CA-altered tumors)
Drug: Letrozole — Letrozole will be administered by mouth once a day on Days 1-28 of each 28-day cycle
  Arms: Inavolisib + Palbociclib + Letrozole (ER+ and PIK3CA-altered tumors)
Drug: Olaparib — Olaparib will be administered by mouth twice a day on Days 1-28 of each 28-day cycle
  Arms: Inavolisib + Olaparib (Non-matched)
Drug: Luteinizing Hormone-Releasing Hormone (LHRH) Agonists — LHRH agonists are required beginning at least 2 weeks prior to initiation of study treatment for premenopausal or perimenopausal women. Acceptable agents include goserelin or leuprolide; triptorelin is also acceptable. Monthly injections of LHRH agonist are preferred.
  Arms: Giredestrant + Abemaciclib (ER+ tumors); Inavolisib + Palbociclib + Letrozole (ER+ and PIK3CA-altered tumors)
Drug: Cyclophosphamide — Cyclophosphamide will be administered by mouth once a day on Days 1-21 of each cycle. (Cycle length = 21 days)
  Arms: Atezolizumab + Bevacizumab + Cyclophosphamide (Non-matched)
Drug: Inavolisib — Inavolisib will be administered by mouth once a day on Days 1-21 of each 21-day cycle
  Arms: Inavolisib + Bevacizumab (PIK3CA-altered tumors)

SUMMARY:
This study will evaluate the efficacy and safety of multiple biomarker-selected treatments in patients with persistent or recurrent rare epithelial ovarian, fallopian tube, or primary peritoneal tumors. Enrollment will take place in two phases: a preliminary phase followed by a potential expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Persistent or recurrent EOC that meets the following criteria: Histologically confirmed non-high-grade serous, non-high-grade endometrioid epithelial ovarian, fallopian tube, or primary peritoneal cancer, including but not limited to low-grade serous ovarian carcinoma, clear cell carcinoma, mucinous carcinoma, carcinosarcoma, undifferentiated carcinoma, seromucinous carcinoma, malignant Brenner tumors, Grades 1 or 2 endometrioid carcinoma, mesonephric-like adenocarcinoma and small cell carcinoma of the ovary, hypercalcemic type (SCCOHT). Disease that is not amenable to curative surgery
* Measurable disease (at least one target lesion) according to RECIST v1.1
* Previous treatment with one to four lines of therapy, at least one of which was platinum-based. Hormonal therapy does not count as a line of therapy.
* Platinum-resistant disease, defined as disease progression during or within 6 months of last platinum therapy, with the following exception: Participants with primary platinum-refractory disease are excluded.
* Submission of a representative tumor specimen that is suitable for next-generation sequencing (NGS) testing and estrogen receptor immunohistochemistry (ER IHC) to determine treatment arm assignment and for central pathology review.
* Submission of the local pathology report and, if available, any associated stained slides that supported the local diagnosis of the histology (to be used for central pathology review)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate hematologic and end-organ function
* For women of childbearing potential: agreement to remain abstinent or use contraception, and agreement to refrain from donating eggs (if applicable)
* In addition to the general inclusion criteria above, participants must meet all of the arm-specific inclusion criteria for the respective arm

General Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant or breastfeed during the study
* Primary platinum-refractory disease, defined as progression during or within 4 weeks after the last dose of the first-line platinum treatment
* Histologic diagnosis of high-grade serous or high-grade endometrioid ovarian, fallopian tube, or primary peritoneal cancer
* Current diagnosis of solely borderline epithelial ovarian tumor
* Current diagnosis of non-epithelial ovarian tumors
* Current diagnosis of synchronous primary endometrial cancer
* Prior history of primary endometrial cancer, with the following exception: a prior diagnosis of primary endometrial cancer is permitted if it meets all of the following conditions: Stage IA, no lymphovascular invasion, International Federation of Gynecology and Obstetrics Grade 1 or 2, not a high-grade subtype.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Symptomatic, untreated, or actively progressing CNS metastases
* Severe infection within 4 weeks prior to initiation of study treatment
* Treatment with chemotherapy, radiotherapy, antibody therapy or other immunotherapy, gene therapy, vaccine therapy, or investigational therapy within 28 days prior to initiation of study treatment
* Treatment with hormonal therapy within 14 days prior to initiation of study treatment
* In addition to the general exclusion criteria above, participants can not meet any of the arm-specific exclusion criteria for the respective arm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 176 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (ORR) | Up to approximately 5 years
  Confirmed ORR is defined as the proportion of participants with a confirmed complete response (CR) or partial response (PR) (demonstrated on two consecutive occasions >=4 weeks apart), as determined by the investigator according to RECIST v1.1.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to approximately 5 years
  DOR is defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1.
Disease Contral Rate (DCR) | Up to approximately 5 years
  DCR is defined as the proportion of participants with a confirmed CR or PR, or stable disease maintained for at least 16 weeks, as determined by the investigator according to RECIST v1.1.
Progression Free Survival (PFS) | Up to approximately 5 years
  PFS after start of treatment is defined as the time from start of treatment to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1.
6-Month PFS Rate | Up to 6 month
  6-month PFS rate is defined as the proportion of participants who remained alive and progression-free at 6 months after start of treatment, as determined by the investigator according to RECIST v1.1.
Overall Survival (OS) | Up to approximately 5 years
  OS after start of treatment is defined as the time from start of treatment to death from any cause.
Confirmed ORR as Determined by IRC (Independent Review Committee) | Up to approximately 5 years
  Confirmed ORR, as determined by the IRC according to RECIST v1.1.
DOR as Determined by IRC | Up to approximately 5 years
  DOR, as determined by the IRC according to RECIST v1.1
DCR as Determined by IRC | Up to approximately 5 years
  DCR, as determined by the IRC according to RECIST v1.1
PFS as Determined by IRC | Up to approximately 5 years
  PFS, as determined by the IRC according to RECIST v1.1
Percentage of Participants With Adverse Events | Up to approximately 5 years
  Percentage of participants with adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (41):
- United States (8):
  - UCSF Helen Diller Family CCC, San Francisco, California
  - Washington University School of Medicine, St Louis, Missouri
  - Levine Cancer Institute, Charlotte, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Texas Oncology - Gulf Coast, The Woodlands, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
- Cabrini Hospital, Malvern, Victoria, Australia
- Canada (2):
  - Princess Margaret Cancer Center, Toronto, Ontario
  - McGill University Health Centre - Glen Site, Montreal, Quebec
- Gynekologicko-porodnicka klinika, Prague, Czechia
- France (8):
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - Centre Francois Baclesse, Caen
  - Centre Leon Berard, Lyon
  - Groupe Hospitalier Diaconesses, Paris
  - Centre Eugène Marquis, Rennes
  - ICO - Site René Gauducheau, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif
- Germany (2):
  - Kliniken Essen-Mitte Evang. Huyssens-Stiftung, Klinik für Gynäkologie und gynäkologische Onkologie, Essen
  - Universitätsklinikum Mannheim, Mannheim
- Italy (4):
  - A.O. U. Consorziale Policlinico di Bari, Bari, Apulia
  - Istituto Tumori Napoli, Napoli, Campania
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - IRCCS S. Raffaele, Milan, Lombardy
- LLC Medscan, Moskva, Moscow Oblast, Russia
- South Korea (4):
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (4):
  - Institutio Catalan De Oncologia, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
- Hôpitaux Universitaires de Genève, Geneva, Switzerland
- Turkey (Türkiye) (3):
  - Adana Baskent University Medical Faculty; Oncology, Adana
  - Baskent Universitesi Ankara Hastanesi; Tıbbi Onkoloji Bölümü, Ankara
  - Koc University Medical Faculty; Department of Gynecology & Obstetrics, Istanbul
- United Kingdom (2):
  - Western General Hospital, Edinburgh
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing